CLINICAL TRIAL: NCT07313826
Title: Neurolumen for Chronic Lower Back Pain: A Pilot RCT Study
Brief Title: Treatment of Chronic Lower Back Pain With a Combination of Electrical Stimulation, LED, and Laser Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Collaborators: Neurolumen LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USUHS.2025-167
Record Dates: First submitted 2025-12-30; First posted 2026-01-02 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low Back Pain
Keywords: chronic pain; low back pain; electrical stimulation; laser therapy
MeSH Terms: conditions — Chronic Pain; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Active Neurolumen device compared to inactive/sham
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Neurolumen (Experimental): The Active Neurolumen group will utilize an active device
  Interventions: Device: Active Neurolumen
- Inactive Neurolumen (Sham Comparator): The Inactive Neurolumen group will utilize an inactive device
  Interventions: Device: Inactive Neurolumen

INTERVENTIONS:
Device: Active Neurolumen — Neurolumen has been cleared by the FDA for the treatment of pain (FDA: 142025) and utilizes a combination of low-level lasers, Light-Emitting Diodes, and electrical stimulation over a 30-minute treatment period to target inflammation and circulation to the affected area. Participants will use the device daily for 4 weeks.
  Arms: Active Neurolumen
Device: Inactive Neurolumen — The sham Neurolumen device will look the same an the Active Neurolumen, and will appear to turn on, but will not provide any treatment
  Arms: Inactive Neurolumen

SUMMARY:
This study will evaluate the impact of the Neurolumen medical device on chronic low back pain.

DETAILED DESCRIPTION:
Chronic low back pain is debilitating and difficult to treat. The commercially-available Neurolumen medical device uses a combination of electrical stimulation, low-level laser, and LED therapies to treat pain. Separately, each of these treatments has shown promise for treating chronic pain. In a recent survey by the manufacturer involving over 4700 Veterans who were prescribed a Neurolumen device through their local VA facility, 93% of patients reported a reduction in pain levels, and 52% report reduction in medication, including 6% who reported cessation of all medication. Additionally, average pain levels of 7.01/10 dropped to 3.38/10 after 6 weeks of use (unpublished data). Thus, there is theoretical support and preliminary evidence for the utility of Neurolumen for treating chronic pain; yet, it is unknown whether these findings generalize to other populations. Furthermore, while a reduction in retrospective pain and medication use are promising, prospectively-collected clinical outcomes of Neurolumen use have yet to be examined. This study will examine the feasibility and efficacy of the Neurolumen devices for treating chronic lower back pain using a double-blind pilot randomized controlled trial design with a placebo/waitlist control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with LBP with an average pain score of 4 or higher on DVPRS for > 3 months
* Ability to sit or lay down for 30 minutes during treatments
* Demonstrated ability to correctly use the device and maintain adequate sensor contact throughout (assisted or unassisted)
* Female participants who could possibly become pregnant must agree to use a highly effective contraceptive method from the screening period through the 4 weeks of study intervention and any use during the wait-list control period. These methods include a physical barrier method (e.g., condom) plus an additional hormonal, IUD, tubal ligation, or second type of barrier (e.g., diaphragm). In addition, they must abstain from egg collection or donation during the same period.

Exclusion Criteria:

* Individuals < 18 or >70 years of age at enrollment
* Persons with Pacemakers, or interstitial pumps, or spinal cord stimulator in ON mode.
* Persons who have received back surgery (open) within the last 3 months
* Pregnant or sexually active female subjects who could possibly become pregnant and who are not willing to use an acceptable form of contraception (barrier method plus one of the following: second barrier, hormonal, IUD, or tubal ligation).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Weeks 1-12
  Defense and Veterans Pain Rating Scale. On a scale of 0-10, with higher scores denoting more pain.
Pain Medication Use | Weeks 1-12
  Opioid Use Diary

SECONDARY OUTCOMES:
Physical Function | Weeks 1-12
  Patient-Reported Outcomes Measurement Information System (PROMIS) -29 Adult Profile 2.0 Instrument, Physical Function subscale.
  Each item is scored on a scale 1-5, with 1=without any difficulty and 5=unable to do. Items will be summed and t-scored (0-100)
Sleep Disturbance | Weeks 1-12
  Patient-Reported Outcomes Measurement Information System (PROMIS) -29 Adult Profile 2.0 Instrument, Sleep Disturbance subscale. Each item is scored on a scale 1-5, with 1=not at all and 5=very much. Items will be summed and t-scored (0-100), with higher scores denoting more sleep disturbance.

OTHER OUTCOMES:
Pain Catastrophizing | Weeks 1-12
  University of Washington Concerns About Pain Six Item Short Form (UW-CAP SF-6). Each item is scored on a scale of 1-5, with 1=never and 5=always. Items are summed and t-scored (0-100), with higher scores denoting more pain catastrophizing.
Perceived Efficacy | Weeks 1-12
  Patient Global Impression of Change Scale (PGIC). Each item is scored on a scale 1-5, with 1=very much improved and 7= Very much worse. Items will be summed and t-scored (0-100), with higher scores denoting more negative change.

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States